CLINICAL TRIAL: NCT02017418
Title: The Effects of a Zeaxanthin Intervention on Visuomotor Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: ZeaVision, LLC (Industry)
Responsible Party: Principal Investigator, Billy R. Hammond, Professor and Principal Investigator, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012-10531
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Behavior and Behavior Mechanisms
Keywords: zeaxanthin; visual function; reaction time; processing speed
MeSH Terms: conditions — Behavior | interventions — Zeaxanthins; Lutein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- zeaxanthin (Experimental): placebo zeaxanthin
  Interventions: Dietary Supplement: zeaxanthin
- combinatory supplement (Active Comparator): placebo combinatory supplement
  Interventions: Dietary Supplement: combinatory supplement

INTERVENTIONS:
Dietary Supplement: zeaxanthin — softgel
  Arms: zeaxanthin
Dietary Supplement: combinatory supplement — softgel
  Other Names: zeaxanthin + lutein + DHA
  Arms: combinatory supplement

SUMMARY:
This study was designed to test whether two zeaxanthin formulations (supplements containing different nutritional compounds with zeaxanthin and omega fatty acids being the primary ingredients of interest) influenced visual motor function. Visual motor function refers to the processing speed of the visual system and how individuals respond behavioral to visual stimuli (e.g., reaction time).

DETAILED DESCRIPTION:
This study was designed to test whether two zeaxanthin formulations (supplements containing different nutritional compounds with zeaxanthin and omega fatty acids being the primary ingredients of interest) influenced visual motor function. Visual motor function refers to the processing speed of the visual system and how individuals respond behavioral to visual stimuli (e.g., reaction time).

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 and ≤ 40 years
* BMI: ≥ 20 and ≤ 30 kg/m2
* No anticipated changes in dieting habits (as relevant to the intake of xanthophylls and fats/oils).
* No anticipated surgical procedures.
* Willingness and ability to give written informed consent and willingness and ability to comply with the study requirements.
* Corrected visual acuity (ETDRS): better than 20/60 in the eye selected for the study

Exclusion Criteria:

* Smokers
* Current or history of relevant ocular diseases (such as AMD) or other conditions e.g., lipid disorders.
* Inability to reliably perform macular pigment optical density measurements by "Heterochromatic Flicker Photometry" or any of the other ophthalmic tests of the study.
* Any condition likely to interfere with normal gastro-intestinal absorption of xanthophylls (e.g., digestive disorders: inflammatory bowel disease, ulcerative colitis, Crohn's, irritable bowel, etc. or lipid disorders including conditions such as hypercholesterolemia)
* Current use of xanthophyll containing supplements or use of xanthophyll containing supplements in the past 6 months (but excluding multivitamins containing lutein or zeaxanthin at low potency).
* Participation in any other study during last 1 month before study initiation.
* Known hypersensitivity or allergy to xanthophylls.
* Regular intake of medications or supplements, which the principal investigator deems likely to confound the study outcomes. These include diabetes medication and statins or any other drug/supplement to modulate cholesterol or fat digestion/absorption.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Macular pigment optical density | one year
  Increases in the amount of macular pigment measured in optical density units

SECONDARY OUTCOMES:
fixed reaction time | one year
  reaction time to a stimulus fixed in space
variable reaction time | 12-months
  reaction time to a stimulus with a position that varies in space
coincidence anticipation | 12-months
  button press when a light stimulus of varying speeds reaches a specific point in a linear light array

CONTACTS AND LOCATIONS:
Overall Officials: Billy R Hammond, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- Department of Psychology, UGA, Athens, Georgia, United States